CLINICAL TRIAL: NCT03991065
Title: Risk of GAstric Adenocarcinoma After Cephalic Duodenopancreatectomy : RAGAD Study
Brief Title: Risk of GAstric Adenocarcinoma After Cephalic Duodenopancreatectomy
Acronym: RAGAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P180302J
Record Dates: First submitted 2019-05-24; First posted 2019-06-19 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Cephalic Duodenopancreatectomy 10 or More Years Ago

STUDY DESIGN:
Intervention Model Description: Of the patients included in the cohort, some will be eligible to perform the endoscopy added for research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with endoscopy (Experimental): high digestive endoscopy
  Interventions: Diagnostic Test: high digestive endoscopy
- without endoscopy (No Intervention): no endoscopy

INTERVENTIONS:
Diagnostic Test: high digestive endoscopy — high digestive endoscopy with biopsies performed according to the sydney protocol
  Arms: with endoscopy

SUMMARY:
In view of the similarities of the surgical set-ups of partial gastrectomies and cephalic duodenopancreatectomies, and the increased risk of gastric cancer after early partial gastrectomy, it is possible that the former pancreatic cephalic duodenopancreatectomy pancreaticoduodenectomy (CPD) is also associated with the occurrence of stomach cancer.

The investigators expect a high rate of cancer and high grade dysplasia in these patients based on literature data and available data on gastric cancer after partial gastrectomy. Participants with lesions to be discovered will benefit from earlier medical management of less advanced tumor lesions, with improved prognosis.

The primary objective of this study is to evaluate the incidence of gastric cancer or high grade dysplasia in patients with old CPP CPD (10 years or older) and who performed the endoscopy protocol.

The cohort will consist of all eligible patients identified from pathology registries and PMSI data from participating centers (patients living 10 years after CPDP, with no previous history of gastric cancer before entering the cohort).

Entry into the cohort (beginning of exposure) will be 10 years after CPD. If a gastric cancer has been diagnosed previously at the beginning of the current study (2019) with histological documentation present in the medical file, no new endoscopy will be performed and the patient will be considered as a "new case" on the date of histological diagnosis of cancer.

Of the patients included in the cohort, some will be eligible to perform the endoscopy added for research. This group will be the sample in which the primary endpoint will be measured.

1. Recruitment of patients with cephalad cephalic duodenopancreatectomy 10 or more years ago 2.

Per patient (in the group with endoscopies):

* Inclusion consultation with patient consent collection
* Anesthesia consultation
* Upper gastrointestinal endoscopy and biopsy
* Follow-up consultation to report the results to the patient and possibly organize a support (announcement device complies with HAS recommendations). For patients in the cohort not included in the endoscopy study, the data collection will be retrospective only (no specific patient consultation for research and no endoscopy review added for this research).

  3. Data analysis: primary endpoints (incidence rate of high grade dysplasia and gastric cancer) and secondary endpoints 700 to 800 patients will be included in the entire cohort and 164 patients in the group with endoscopy.

  7 centers in Ile de France participate.
* duration of inclusion: 36 months
* duration of participation (treatment + follow-up): schedule of the visit of anesthesia (5.5 months max), endoscopy programming (1 month max) + the day of the exam + 4 weeks for the results of the exam: 8 months maximum
* total duration: 44 months

DETAILED DESCRIPTION:
In view of the similarities of the surgical set-ups of partial gastrectomies and cephalic duodenopancreatectomies, and the increased risk of gastric cancer after early partial gastrectomy, it is possible that the former pancreatic cephalic duodenopancreatectomy (CPD) is also associated with the occurrence of stomach cancer.

The investigators expect a high rate of cancer and high grade dysplasia in these patients based on literature data and available data on gastric cancer after partial gastrectomy. Participants with lesions to be discovered will benefit from earlier medical management of less advanced tumor lesions, with improved prognosis.

The investigators results will provide an argument for conducting larger analytical studies and will also provide useful information for the design of these studies. These studies will eventually identify a gastric cancer screening strategy among patients with previous CPDP. Screening programs in groups at higher risk of gastric cancer among patients with CPDP could provide significant benefits in terms of gastric cancer mortality and quality of life, as well as medico-economic positive for the health care system.

The primary objective of this study is to evaluate the incidence of gastric cancer or high grade dysplasia in patients with old CPDP (10 years or older) and who performed the endoscopy protocol.

The primary endpoint is the incidence rate of gastric cancer or high grade dysplasia in patients who had CPDP 10 years or more ago.

The cohort will consist of all eligible patients identified from pathology registries and PMSI data from participating centers (patients living 10 years after CPDP, with no previous history of gastric cancer before entering the cohort).

Entry into the cohort (beginning of exposure) will be 10 years after CPD. If a gastric cancer has been diagnosed previously at the beginning of the current study (2019) with histological documentation present in the medical file, no new endoscopy will be performed and the patient will be considered as a "new case" on the date of histological diagnosis of cancer. The collection of data will be retrospective for these patients.

Of the patients included in the cohort, some will be eligible to perform the endoscopy added for research. This group will be the sample in which the primary endpoint will be measured.

1. Recruitment of patients with cephalad cephalic duodenopancreatectomy 10 or more years ago 2.

Per patient (in the group with endoscopies):

* Inclusion consultation with patient consent collection
* Anesthesia consultation
* Upper gastrointestinal endoscopy and biopsy
* Follow-up consultation to report the results to the patient and possibly organize a support (announcement device complies with HAS recommendations). For patients in the cohort not included in the endoscopy study, the data collection will be retrospective only (no specific patient consultation for research and no endoscopy review added for this research).

  3. Data analysis: primary endpoints (incidence rate of high grade dysplasia and gastric cancer) and secondary endpoints 700 to 800 patients will be included in the entire cohort and 164 patients in the group with endoscopy.

  7 centers in Ile de France participate.
* duration of inclusion: 36 months
* duration of participation (treatment + follow-up): schedule of the visit of anesthesia (5.5 months max), endoscopy programming (1 month max) + the day of the exam + 4 weeks for the results of the exam: 8 months maximum
* total duration: 44 months

ELIGIBILITY:
1. Inclusion Criteria:

   Criteria for inclusion for patient without endoscopy for research:
   * Patient living 10 years after a CPD performed for a benign or malignant condition in one of the participating centers
   * Age ≥ 18 years at the time of entry into the cohort (10 years after CPD)
   * Non opposition to the use of data
   * patient with endoscopy realised 10 years after CPD and before the participation of the study

   Inclusion criteria to have endoscopy :
   * Patient living 10 years after a CPP performed for a benign or malignant condition in one of the participating centers Age ≥ 18 years of age for inclusion in the "endoscopy" group
   * Patient with low or medium anesthetic risk (ASA 1, ASA 2, ASA 3)
   * Patient who does not have a genetic or acquired haemostasis disorder preventing the performance of gastric biopsies
   * Possibility of stopping treatment with anticoagulant or clopidogrel or ticagrelor if necessary (see Appendix 1: Management of anticoagulants-antiaggregants in upper gastrointestinal endoscopy requiring gastric biopsies (according to SFED, ESGE recommendation)) (44)
   * Patient affiliated to a social security scheme
   * Informed and signed consent of the patient obtained
2. No inclusion Criteria:

Criteria for non-inclusion for all patient:

- Personal history of gastric cancer prior to inclusion in the cohort (before CPD or 10 years after CPD)

Criteria for non-inclusion in endoscopy'group:

* Personal history of gastric cancer
* Pregnant or lactating woman
* Patient under guardianship
* Patient with contraindications to local anesthetics and propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
the incidence rate of gastric cancer or high grade dysplasia in patients who had CPD 10 or more years ago in the sample of patients who performed the protocol endoscopy | 7 months after inclusion
  the ratio of the number of new cases of gastric cancer or high grade dysplasia (diagnosed at endoscopy with biopsies) divided by the sum of person-times at risk of developing the disease (expressed in person-years).

SECONDARY OUTCOMES:
Prevalence of gastric cancer or high grade dysplasia in patients who performed the endoscopy | 7 months after inclusion
  the proportion of patients with gastric cancer or high grade dysplasia among patients in the endoscopic study
Low-grade dysplasia incidence rate in patients who performed the endoscopy | 7 months after inclusion
  ratio of the number of new cases of low-grade dysplasia (diagnosed at endoscopy with biopsies) divided by the sum of person-times at risk of developing the disease ( expressed in person-years)
prevalence of low grade dysplasia in patients who performed the endoscopy | 7 months after inclusion
  proportion of patients with low grade dysplasia
Incidence rate of intestinal metaplasia in patients who performed the endoscopy | 7 months after inclusion
  ratio of the number of new cases of intestinal metaplasia (diagnosed at endoscopy with biopsies) divided by the sum of person-times at risk of developing the disease (expressed in terms of years)
prevalence of intestinal metaplasi in patients who performed the endoscopy | 7 months after inclusion
  proportion of patients with intestinal metaplasia.
incidence rate of gastric cancer or high grade dysplasia in cohort of patients | inclusion
  ratio of the number of new cases of low grade dysplasia (histological evidence in the medical file or diagnosed at the endoscopy provided for in the protocol) divided by the sum of person-times at risk of developing the disease (expressed in person-years)
prevalence of gastric cancer or high grade dysplasia in cohort of patients | inclusion
  proportion of patients with gastric cancer or high grade dysplasia
incidence rate of low-grade dysplasia in cohort of patients | inclusion
  the ratio of the number of new cases of low-grade dysplasia (histological evidence in the medical file or diagnosed at the protocol endoscopy) divided by the sum of the time at risk of developing the disease (expressed in person-years)
prevalence of low grade dysplasia in cohort of patients | inclusion
  proportion of patients with intestinal metaplasia
incidence rate of intestinal metaplasia in cohort of patients | inclusion
  ratio of the number of new cases of low grade dysplasia (histological evidence in the medical file or diagnosed at the endoscopy provided for in the protocol) divided by the sum of the person-times at risk of developing the disease (expressed in person-years)
Prevalence of intestinal metaplasia, in cohort of patients | inclusion
  proportion of patients with intestinal metaplasia factors associated with gastric cancer or severe dysplasia. The factors thought to be associated are: family history of gastric cancer, active smoking, presence of Helicobacter pylori, digestive symptoms, pancreaticogastric anastomosis.
Factors associated with low-grade dysplasia or intestinal metaplasia in cohort of patients | inclusion
  occurence of factors thought to be associated, as well as those of gastric cancer or high-grade dysplasia.

CONTACTS AND LOCATIONS:
Locations (1):
- LORENZO, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided